CLINICAL TRIAL: NCT05131438
Title: An Expanded Access Program to Provide Sugemalimab for the Treatment of Relapsed or Refractory Extranodal Natural Killer/T-Cell Lymphoma (R/R ENKTL)
Status: No longer available | Type: Expanded Access
Sponsor: EQRx International, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: EQ165-501
Record Dates: First submitted 2021-11-11; First posted 2021-11-23 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Extranodal NK/T-cell Lymphoma
Keywords: relapsed/refractory
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Recurrence | interventions — sugemalimab

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: sugemalimab — sugemalimab (Anti-PD-L1 antibody)

SUMMARY:
This program is intended to provide access to sugemalimab for participants with R/R ENKTL, after their disease failed to respond to prior treatment regimen(s), preceding marketing authorization by the local regulatory agency.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to receive sugemalimab as part of this EAP only if all the following criteria apply:

1. Participants must be 18 to 99 years of age inclusive, at the time of signing the informed consent.
2. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
3. Participants who have a histologically confirmed ENKTL. Both nasal and non-nasal ENKTL are allowed.
4. Participants must have R/R ENKTL that has progressed on or after asparaginase-based chemotherapy or chemoradiotherapy. (Relapse: disease progression after response to the last treatment; refractory: no response to the last treatment).
5. Women of childbearing potential (WOCBP), as defined in Section 13.3 must have a negative serum pregnancy test ≤7 days before the first dose of sugemalimab. WOCBP or fertile men and their WOCBP partners must agree to use an effective contraceptive method from providing signed ICF through 6 months after the last dose of the sugemalimab.
6. Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

Participants are not eligible to participate in the Sugemalimab ENKTL EAP if any of the following criteria apply:

1. Participants with aggressive natural killer cell leukemia or ENKTL participants who have any degree of leukemic involvement.
2. Participants with hemophagocytic lymphohistiocytosis.
3. Subjects requiring systemic corticosteroid or any other immunosuppressive therapy. (Subjects are permitted to use topical, ocular, intra-articular, intranasal and inhaled corticosteroids [with minimal systemic absorption]; a short course [≤ 7 days] of corticosteroids for prophylaxis [e.g., hypersensitivity to contrast media] or for treatment of non-autoimmune conditions [e.g., delayed hypersensitivity caused by contacting allergens])
4. Participants with underlying condition that in the treating physician's opinion would increase the risk of AEs related to sugemalimab administration or confound the assessment for its toxicity. Participants who have had prior chemotherapy, immunotherapy, biological therapy (including cancer vaccine, cytokine therapy or growth factors to treat cancer) used as a systemic treatment for cancer will require 28 days of washout period.
5. Participants with active, known or suspected autoimmune disease.
6. Any liver function panel analyte (LFT) value > 2.5 × upper limits of normal reference range (ULN) which includes aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase, and gamma-glutamyl transferase (GGT) at baseline. Bilirubin > 1.5 × ULN.
7. Any positive test for hepatitis B virus or hepatitis C virus indicating acute or chronic infection.
8. Participants in the treating physician's opinion are not suitable for participating in this EAP.

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States